CLINICAL TRIAL: NCT01286142
Title: A Prospective, Observational Safety Study in Children <= 24 Months of Age Receiving Oseltamivir for the Treatment or Prophylaxis of Influenza Infection
Brief Title: Oseltamivir Infant Influenza Safety Study
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Barbara Rath, Principle Investigator, Pediatric Infectious Diseases & Vaccines, Charite University, Berlin, Germany
Other Study IDs: NV25182
Record Dates: First submitted 2011-01-24; First posted 2011-01-31 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Influenza, Human
Keywords: Prospective, Observational Safety Study
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Influenza treatment with oseltamivir: Patients 24 months of age and younger initially presenting with confirmed or presumed influenza A or B infection treated with oseltamivir.
- Influenza prophylaxis with oseltamivir: Patients 24 months of age and younger prescribed oseltamivir for influenza prophylaxis
- Influenza patients with no antiviral treatment: A comparator group of patients 24 months of age and younger presenting with confirmed or presumed influenza A or B and not treated with any influenza antiviral.

SUMMARY:
In June 2009, the World Health Organization (WHO) declared a global pandemic of influenza A (H1N1). Although little is known about the pandemic influenza strain in children, during previous pandemics and influenza seasons children less than one year of age were shown to be at higher risk of influenza complications than older children. In light of the 2009 H1N1 pandemic situation, the U.S. Food and Drug Administration (FDA), European Medicines Agency (EMA), and Health Canada issued emergency authorizations for oseltamivir to be used to treat and prevent influenza in infants under 1 year of age. It is anticipated that oseltamivir use in infants will dramatically increase due to the new authorizations for use in this population and high prevalence of H1N1 influenza circulating in the population. Ongoing safety surveillance is critical and this study will provide further data for evaluating the risk/benefit ratio of prescribing oseltamivir to this population in the current milieu of both seasonal and pandemic influenza viruses circulating in the population. The study will also provide useful information on the dose and duration of treatment used in clinical practice and their relationship to adverse events.

DETAILED DESCRIPTION:
This study is a prospective, observational, multicenter short-term safety study of the use of oseltamivir (prophylaxis or treatment) in children 24 months of age or younger. An internal comparator group of children diagnosed with influenza and not treated with antiviral medications will be enrolled. The study includes a 30-day follow-up period and will be conducted in multiple sites in multiple countries within the European Union. The study will cover two consecutive influenza seasons: 01 October 2009 - 31 May 2010 and 01 October 2010 - 31 May 2011. Data collection may be interrupted in the interim period between influenza seasons (June 1, 2010 - September 30, 2010), depending on whether the influenza season follows the expected cycle.

ELIGIBILITY:
Inclusion Criteria:

* 24 months of age or younger at time of enrollment
* Diagnosis of influenza A or B (suspected* or confirmed by viral testing) either treated with oseltamivir or with no antivirals OR prescribed oseltamivir for post-exposure influenza prophylaxis
* Parent/legal guardian willing to provide informed consent and be contacted by telephone as part of follow-up

Exclusion Criteria:

* Patients will be excluded if treated with an influenza antiviral other than oseltamivir, including amantadine, rimantadine, or zanamivir.

  * Suspected influenza is defined as an acute febrile illness characterized by the presence of fever and 1 or more of the following symptoms: cough, coryza/nasal congestion or sore throat.

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study will be conducted in multiple sites in multiple countries within the European Union. Initially, five countries (United Kingdom, Austria, Finland, Poland, Germany) are selected for inclusion, but additional countries in Europe, are likely to be added. It is estimated that 3-12 sites per country will be enrolled, with a target of at least 900 patients. If additional countries are added, the number of sites/patients recruited per country will be adjusted accordingly.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events | Study Day 7 post-baseline
  Information on the number of subjects with AEs will be collected at 7 days post-baseline. AEs include influenza symptoms and associated complications solicited from parent/legal guardian; secondary complications of influenza reported by physician, including otitis media and bacterial infections; and any other non-serious and serious AEs.
Number of subjects with Adverse Events | Study Day 30 post-baseline
  Information on the number of subjects with AEs will be collected at 30 days post-baseline. AEs include influenza symptoms and associated complications solicited from parent/legal guardian; secondary complications of influenza reported by physician, including otitis media and bacterial infections; and any other non-serious and serious AEs.

SECONDARY OUTCOMES:
Number of subjects treated with oseltamivir | Day 30 post baseline
  Data on dosage and duration of treatment with oseltamivir in real-world practice are collected. The aim is to examine the relationship of adverse events to the regimen of oseltamivir.
Number of subjects with drug-resistant virus | Day 30 post-baseline
  Data on oseltamivir resistance are collected (as reported only)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Rath, MD, Principal Investigator — Charite University Berlin, Department of Pediatrics (Div. of Pneumonology and Immunology)
Locations (1):
- Charite University Berlin, Berlin, Germany

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Interim Guidance for Clinicians on the Prevention and Treatment of Novel Influenza A (H1N1) Influenza Virus Infection in Infants and Children. 13 May 2009. Available at http://cdc.gov/h1n1flu/childrentreatment.htm. Accessed 03 Aug 2009.
- [Background] European Medicines Agency (EMA), Committee for Medicinal Products for Human Use. CHMP ASSESSMENT REPORT on Novel Influenza (H1N1) outbreak Tamiflu (oseltamivir) Relenza (zanamivir) [EMEA/CHMP/287662/2009]. 07 May 2009. Available at http://www.emea.europa.eu/humandocs/PDFs/EPAR/tamiflu/28766209en.pdf. Accessed 28 July 2009.
- [Background] Food and Drug Administration (FDA). Emergency Use Authorization Letter - Tamiflu. 14 July 2009. Available at http://www.cdc.gov/h1n1flu/eua/pdf/fda_letter_tamiflu.pdf. Accessed 03 Aug 2009.
- [Background] World Health Organization. 11 Jun 2009. Available at: http://www.who.int/mediacentre/news/statements/2009/h1n1_pandemic_phase6_20090611/en/index.html. Accessed 03 Aug 2009.
- [Background] Centers for Disease Control and Prevention (CDC). Neurologic complications associated with novel influenza A (H1N1) virus infection in children - Dallas, Texas, May 2009. MMWR Morb Mortal Wkly Rep. 2009 Jul 24;58(28):773-8. PMID 19629027
- [Background] Tamura D, Miura T, Kikuchi Y. Oseltamivir phosphate in infants under 1 year of age with influenza infection. Pediatr Int. 2005 Aug;47(4):484. doi: 10.1111/j.1442-200x.2005.02088.x. No abstract available. PMID 16091087
- [Background] Okamoto S, Kamiya I, Kishida K, Shimakawa T, Fukui T, Morimoto T. Experience with oseltamivir for infants younger than 1 year old in Japan. Pediatr Infect Dis J. 2005 Jun;24(6):575-6. doi: 10.1097/01.inf.0000164799.33635.fe. No abstract available. PMID 15933579